CLINICAL TRIAL: NCT04930653
Title: A Phase II Study of Combination Extracorporeal Photopheresis (ECP) and Mogamulizumab in Erythrodermic CTCL
Brief Title: Extracorporeal Photopheresis and Mogamulizumab for the Treatment of Erythrodermic Cutaneous T Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20724; NCI-2021-03533 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20724 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Folliculotropic Mycosis Fungoides; Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Sezary Syndrome; Stage IB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage II Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIA Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IIB Mycosis Fungoides and Sezary Syndrome AJCC v8; Transformed Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides | interventions — Photopheresis; mogamulizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ECP, mogamulizumab) (Experimental): Patients receive mogamulizumab IV over 60 minutes on days 1, 8, 15, 22, of cycle 1 and days 1 and 15 of subsequent cycles. Beginning in cycle 2, patients also undergo ECP over 3 hours on days 8, 9, 22,and 23. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving CR)/PR after 6 cycles receive up to 6 additional cycles of treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Extracorporeal Photopheresis; Biological: Mogamulizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — Undergo ECP
  Other Names: Extracorporeal Photophoresis; photopheresis; Photophoresis
Biological: Mogamulizumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(CC Chemokine Receptor CCR4) (Human-Mouse Monoclonal KW-0761 Heavy Chain), Disulfide With Human-Mouse Monoclonal KW-0761 Kappa-Chain, Dimer; KM8761; KW-0761; Mogamulizumab-kpkc; Poteligeo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of extracorporeal photopheresis (ECP) and mogamulizumab in treating patients with erythrodermic cutaneous T cell lymphoma (CTCL), a type of skin lymphoma. CTCL is a rare type of cancer that begins in the white blood cells called T cells. Erythrodermic is a widespread red rash that may cover most of the body. ECP is a medical treatment that removes blood with a machine, isolates white blood cells and exposes them to ultra violet light, then returns the cells to the body. Mogamulizumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving mogamulizumab with ECP may work together to kill the tumor cells directly (with mogamulizumab) and boost immune response to cancer (with ECP).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess tolerability and overall response rate (ORR) of the (ECP)/mogamulizumab regimen in CTCL patients previously untreated with mogamulizumab.

SECONDARY OBJECTIVES:

I. To estimate complete response (CR) rate, time to response, duration of response, progression free survival, and overall survival in CTCL patients treated with the ECP/mogamulizumab combination.

II. To summarize the toxicities in CTCL patients treated with the ECP/mogamulizumab combination.

EXPLORATORY OBJECTIVES:

I. To assess quality of life (QoL) parameters before, during, and after the regimen.

II. To evaluate the anti-tumor and immunomodulatory effects of mogamulizumab in the CTCL microenvironment in skin and blood samples of erythrodermic CTCL patients.

III. To evaluate the immunomodulatory effects of ECP.

OUTLINE:

Patients receive mogamulizumab intravenously (IV) over 60 minutes on days 1, 8, 15, 22, of cycle 1 and days 1 and 15 of subsequent cycles. Beginning in cycle 2, patients also undergo ECP over 3 hours on days 8, 9, 22,and 23. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR)/partial response (PR) after 6 cycles receive up to 6 additional cycles of treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guideline
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed mycosis fungoides (MF) or Sezary syndrome (SS). Safety lead-in: >= stage IIB OR >= stage IB-IIA folliculotropic/transformed MF. Phase 2: >= stage IB

  * Stage of disease according to Tumor-Node-Metastasis-Blood (TNMB) classification
  * Pathology report must be diagnostic or be consistent with MF/SS criteria
  * SS is defined as meeting T4 plus B2 criteria; where the biopsy of erythrodermic skin may only reveal suggestive but not diagnostic histopathologic features, the diagnosis may be based on either node biopsy or fulfillment of B2 criteria
  * For MF where the histological diagnosis by light microscopic examination is not confirmed, diagnostic criteria that been recommended by the International Society of Cutaneous Lymphomas (ISCL) should be used.
* Measurable disease per Modified Severity Weighted Assessment Tool (mSWAT) and/or Sezary count
* Baseline skin biopsy taken within 6 months available for central review submission
* Without bone marrow involvement: Absolute neutrophil count (ANC) >= 1,500/mm^3 (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: ANC >= 1,000/mm^3 (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Without bone marrow involvement: Platelets >= 100,000/mm^3 (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: Platelets >= 75,000/mm3 (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease)(performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (unless has Gilbert's disease)(performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (unless has Gilbert's disease)(performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (unless has Gilbert's disease) (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Hepatitis C virus (HCV)*, active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Subjects with MF and a history of staphylococcus colonization are eligible provided they continue to receive stable doses of prophylactic antibiotics
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior mogamulizumab
* Any systemic therapy, including monoclonal antibody within 28 days or 5 half-lives (whichever is shorter) of initiating protocol therapy
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy
* Any skin-directed therapy within 14 days prior to initiating protocol therapy
* Any radiation therapy within 21 days prior to initiating protocol therapy
* Immunosuppressive medication within 14 days prior to the first dose of study treatment. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection) and are on stable dose for at least 28 days
  * Systemic corticosteroids at physiologic doses of < 10 mg/day of prednisone or equivalent
* Live, attenuated vaccine within 30 days prior to the first dose protocol therapy
* Disease free of prior malignancies for >= 5 years with the exception of:

  * Currently treated squamous cell and basal cell carcinoma of the skin, or
  * Carcinoma in situ of the cervix, or
  * Surgically removed melanoma in situ of the skin (stage 0) with histological confirmed free margins of excision, or
  * Prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) that has/have been surgically cured, or
  * Any other malignancy that has/have been curatively treated with surgery and/or localized radiation
* Active infection requiring antibiotics
* Known hepatitis B or hepatitis C infection
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Prior stem cell transplantation
* Acute infection requiring systemic treatment
* Conditions requiring chronic steroid or immunosuppressive treatment that likely need additional steroid or immunosuppressive treatments in addition to the protocol therapy
* Renal failure requiring hemodialysis or peritoneal dialysis
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* Major surgery (as defined by the investigator) within the 28 days prior to the first dose of study treatment
* Active or prior documented autoimmune or inflammatory disorders requiring therapy within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Vitiligo or alopecia
  * Hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; or
  * Psoriasis not requiring systemic treatment
* History of primary immunodeficiency
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year post treatment
  ORR will be calculated as the proportion of evaluable patients that have confirmed complete response (CR) or partial response (PR), as defined according to global response assessment. Exact 95% confidence intervals will be calculated for these estimates.
Incidence of adverse events | Up to cycle 3 (each cycle = 28 days)
  Toxicity and adverse events will be recorded using the National Cancer Institute Common Terminology Criteria for Adverse Events 5.0 scale. Observed toxicities will be summarized by type, severity, date of onset, and attribution.

SECONDARY OUTCOMES:
Complete response rate | Up to 1 year post treatment
  Defined as the proportion of response-evaluable patients that have a documented CR.
Time to response | From initiation of study therapy to the first achievement of CR or PR, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Duration of response | From the first achievement of PR or CR to time of partial disease or death, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Progression-free survival | From initiation of study therapy to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival | From initiation of study therapy to death from any cause, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Incidence of adverse events | Up to 30 days post treatment
  Toxicity and adverse events will be recorded using the National Cancer Institute Common Terminology Criteria for Adverse Events 5.0 scale. Observed toxicities will be summarized by type, severity, date of onset, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane R Querfeld, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia